CLINICAL TRIAL: NCT05008874
Title: Prospective, Retrospective, Multicenter, Observational Study of Disease Progression in Adults With Inherited Forms of Spastic Paraplegia
Brief Title: Study of Disease Progression in Adults With Inherited Forms of Spastic Paraplegia
Acronym: CYGNET
Status: Terminated | Type: Observational
Why Stopped: The AMN program requires significantly more time, patients, and resources, including the manufacture of additional investigational product, than what is currently available to Spur.
Sponsor: SwanBio Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: SBTNHX-CT901
Record Dates: First submitted 2021-08-12; First posted 2021-08-17 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-06

CONDITIONS: AMN; AMN Gene Mutation; X-ALD
Keywords: AMN; X-ALD; Natural History; Adrenoleukodystrophy; X-linked Adrenoleukodystrophy; Adrenomyeloneuropathy; Myeloneuropathy; Spastic paraplegia; Hereditary Spastic Paraplegia; HSP; ALD; ABCD1; ALDP; CALD; CCALD; Brain Diseases, Metabolic, Inborn; Brain Diseases, Metabolic; Hereditary Central Nervous System Demyelinating Diseases; Leukoencephalopathies; Demyelinating Diseases; Heredodegenerative Disorders, Nervous System; Metabolism, Inborn Errors; Peroxisomal Disorders; Metabolic Diseases; Adrenal Insufficiency
MeSH Terms: conditions — Adrenoleukodystrophy; Paraplegia; Spastic Paraplegia, Hereditary; Brain Diseases, Metabolic, Inborn; Brain Diseases, Metabolic; Hereditary Central Nervous System Demyelinating Diseases; Leukoencephalopathies; Demyelinating Diseases; Heredodegenerative Disorders, Nervous System; Metabolism, Inborn Errors; Peroxisomal Disorders; Metabolic Diseases; Adrenal Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Males with AMN: Adult males with confirmed diagnosis of ALD and symptoms of AMN.
  Interventions: Other: Natural History Observation

INTERVENTIONS:
Other: Natural History Observation — Data collection on progression of disease

SUMMARY:
The course of AMN-related disabilities over time is poorly or incompletely understood due to a limited number of patients and lack of treatments. This study will help obtain a better understanding of the progression of disease with AMN and facilitate efficient clinical development of future interventional medications.

DETAILED DESCRIPTION:
Progressive weakness and spasticity of the legs are characteristics of numerous disorders and conditions, including those that are inherited neurological disorders.

Adrenomyeloneuropathy (AMN) is an example of an inherited form of spastic paraplegia.

Adrenoleukodystrophy (ALD) is a progressive neurodegenerative disorder caused by a mutation in the ABCD1 gene localized to the X-chromosome (Xq28). The ABCD1 gene encodes a peroxisomal adenosine triphosphate (ATP) binding cassette transporter responsible for transport of very long chain fatty acids (VLCFA) from the cytosol into the peroxisome for degradation. A mutation in ABCD1 results in reduction in the degradation of the VLCFA by peroxisomal β-oxidation, and saturated VLCFA, in particular C26:0, accumulate in tissues and body fluids (i.e., brain, nervous system, adrenal glands). One of the key clinical symptoms during aging of ALD patients is a slowly progressive axonopathy affecting sensory ascending and motor descending spinal cord tracts with 100% penetrance in men, an ALD phenotype known as AMN. There are no treatment options available, which leaves AMN patients with a progressive disorder that leads to lifelong physical disability. The progressive dying-back axonopathy represents the core clinical feature of AMN, with onset usually between 20 and 30 years of age in male participants. The initial symptoms include progressive stiffness and weakness of the legs, impaired vibration and position senses in the lower limbs, falls, sphincter disturbances and impotence, as well as scarce scalp hair (alopecia). About 66% of male AMN patients have adrenocortical insufficiency (Addison disease).

The course of AMN-related disabilities over time is poorly or incompletely understood due to a limited number of patients and lack of treatments. This study will help obtain a better understanding of the progression of disease with AMN and facilitate efficient clinical development of future SwanBio interventional medications.

ELIGIBILITY:
Inclusion Criteria:

1. Male adults aged ≥18 years
2. Diagnosed with ALD based on elevated VLCFA assay and pedigree analysis
3. Clinical evidence of spinal cord involvement with EDSS score between 1 and 6.5

Exclusion Criteria:

1. Diagnosed with cerebral inflammatory disease or has a history of diagnosis with cerebral inflammatory disease
2. Unstable, clinically significant neurologic (other than the disease being studied), psychiatric, cardiovascular, ophthalmologic, pulmonary, hepatic, renal, metabolic, gastrointestinal, urologic, immunologic, hematopoietic, or endocrine disease (other than adrenal insufficiency) or other abnormality, which may impact the ability to participate in the study or that may potentially confound the study results
3. Participant who, in the opinion of the Investigator, has any other medical or psychological condition or social circumstances which would impair their ability to participate reliably in the assessments, or who may increase the risk to themselves or others by participating

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult males diagnosed with ALD (without cerebral disease) and symptoms of AMN who have no other major confounding comorbidities.
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2021-06-21 (Actual); Primary Completion 2025-05-16 (Actual); Study Completion 2025-05-16 (Actual)

PRIMARY OUTCOMES:
Disease progression | 5 years
  Characterize disease progression in adults diagnosed with AMN in serial clinical evaluations of walking

SECONDARY OUTCOMES:
Change in Quality of Life | 5 years
  Characterize the Change in multiple Quality of Life (QoL) parameters over time

CONTACTS AND LOCATIONS:
Locations (6):
- United States (4):
  - Stanford Neuroscience Health Center, Stanford, California
  - Massachusetts General Hospital, Boston, Massachusetts
  - Weill Medical College of Cornell University, New York, New York
  - University of Utah, Salt Lake City, Utah
- University of Leipzig Medical Center, Leipzig, Germany
- Amsterdam UMC, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided